CLINICAL TRIAL: NCT02909608
Title: Investigation of Actigraphy, an Exercise Measurement Device, as a Novel, Well-defined, Reliable, Feasible, Easy to Use, and Non-Invasive Study Endpoint to Facilitate Pediatric Pulmonary Arterial Hypertension Trials and Drug Development
Brief Title: Actigraphy in Pediatric Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1422
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls
  Interventions: Other: No interventions / observations only
- Children With Pulmonary Hypertension
  Interventions: Other: No interventions / observations only

INTERVENTIONS:
Other: No interventions / observations only — This is an observational study only
  Other Names: There are no interventions as part of this study

SUMMARY:
Physical activity is an important factor in understanding how diseases can affect a child. Decreases in physical activity are sometimes the first thing that happens before a child is diagnosed with a disease. When a child sees their doctor, that visit reflects a single point in time. It does not capture how a child feels during the days in between visits to their doctor. This study plans to use special monitors called actigraphs to collect information about physical activity in children with a type of disease called pulmonary hypertension. This study will measure how active these children are and compare their activity to clinical information and to actigraphy measurements in children without pulmonary hypertension.

DETAILED DESCRIPTION:
Pediatric pulmonary arterial hypertension (PAH) (roughly 1-5 cases per 1 million children) is a severe disorder with high mortality and morbidity, but limited treatment options. Pediatric PAH is defined the same as that in adults, which is the presence of abnormally high pulmonary artery pressure. In comparison with adults, pediatric PAH is likely a more severe disorder with higher mortality and morbidity without treatment. Except for INOmax for persistent pulmonary hypertension of the newborn, no drug is currently approved in the US to treat pediatric PAH patients 1-17 years of age. Drug development to treat pediatric PAH is an unmet public health need for children and a priority for the Food and Drug Administration (FDA). However, studies that address the safety and efficacy of PAH therapies are rare, in part due to the lack of suitable clinical endpoints and quantitative and qualitative measures of disease severity.

A major limitation towards enhancing outcomes of children with PAH is the lack of pediatric efficacy endpoints or surrogate measures that are capable of reproducibly and reliably reflecting changes in pulmonary arterial pressure in response to a therapeutic intervention that is being assessed in a pediatric clinical trial. Children are often too young and developmentally unable to perform standard cardiopulmonary exercise testing and the use of several metrics are not as accurate for reflecting clinical status in children as in adults, such as 6 minute walking distance. Additionally, the use of cardiac catheterization to directly measure pulmonary vascular resistance is invasive, requires anesthesia, and has additional risks for complications.

Therefore, to address this critical and unmet medical need in children with PAH, we propose to begin develop a novel, developmentally-appropriate non-invasive endpoint in children through the use of actigraphy. Actigraphy is a mobile device that directly, reproducibly and non-invasively measures physical activity, which can be readily assessed in the ambulatory setting, and may provide a novel, simple and inexpensive approach. Impaired exercise tolerance is a prominent feature of PAH and contributes significantly to reduced quality of life. Assessing exercise capacity is an integral part of the clinical evaluation of PAH in adults and the use of the 6 minute walk distance (6MWD) is the most common primary endpoint in adult PAH clinical trials. Importantly, the 6MWD test and other existing exercise performance tests that are readily applied in adult studies are not reliable and applicable for young children and infants. We propose that actigraphy may provide a novel endpoint for assessing drug efficacy in children if proven to be strongly predictive and reflect clinical course and outcomes of children with PAH. If successful, this early study has great potential for having a significant regulatory impact that will advance the public health mission, as actigraphy could possibly become an endpoint that would be accepted in pediatrics as a regulatory standard for PAH clinical trials.

The purpose of the current study is to describe the use of actigraphy in children with PAH and to determine if correlations exist between actigraphy data and clinical data in children with PAH.

ELIGIBILITY:
Inclusion Criteria for children with PAH:

1. Ages 8-14 years at the time of consent
2. Current diagnosis of pulmonary hypertension in WHO Diagnostic Group 1 as per established clinical criteria

Inclusion Criteria for Control children:

1. Ages 8-14 years at the time of consent
2. Absence of significant cardiopulmonary disease as per medical history

Exclusion criteria for children with PAH:

1. Current disease severity of Panama functional class IIIb or IV
2. Any bone, neuromuscular, or other pathology that may limit activity
3. Use of any medications known to limit activity
4. Active infection, or has any of the following:

   * cardiovascular,
   * liver,
   * renal,
   * hematologic,
   * gastrointestinal,
   * immunologic,
   * endocrine,
   * metabolic, or
   * central nervous system

   disease or condition that, in the opinion of the Investigator, may adversely affect the safety of the subject or interfere with the interpretation of study assessments.
5. Actively listed for transplantation
6. Subject and/or legal guardian has/have

   * an unstable psychiatric condition or
   * is/are mentally incapable of understanding the objectives, nature, or consequences of the trial, or
   * has any condition in which the Investigator's opinion would constitute an unacceptable risk to the subject's safety.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will include children with pulmonary hypertension and children without pulmonary hypertension into this study. All enrolled children must be between the ages of 8-14 years at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Investigate and define the utility of the measurement properties of actigraphy in children with PAH: Baseline | Baseline
  Children will wear both actigraphy devices for 2 weeks at 2 different time points. The first time point is at Baseline when the child enters the study. The second time point is at Week 26, which is 26 weeks after the Baseline timepoint.
Investigate and define the utility of the measurement properties of actigraphy in children with PAH: Week 26 | Week 26
  Children will wear both actigraphy devices for 2 weeks at 2 different time points. The first time point is at Baseline when the child enters the study. The second time point is at Week 26, which is 26 weeks after the Baseline timepoint.

SECONDARY OUTCOMES:
Use statistical analysis to determine correlations of actigraphy with disease severity, progression, clinical worsening, and survival, based on data from this prospective clinical study. | For 18 months
  Children with PH will have information collected from their medical charts that will be compared to their actigraphy data

CONTACTS AND LOCATIONS:
Overall Officials: Dunbar Ivy, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleppinger C, Ivy D, Stockbridge N, Bates A, Handler S, Krishnan US, Mullen MP, Yung D, Hopper RK, Varghese NP, Fineman J, Austin ED, Avitabile CM, Freire G, Clark J, Sun H. Procedural Variation May Contribute to 6-Minute Walk Distance Variability in Real-World Pediatric Pulmonary Arterial Hypertension Study. AAPS J. 2025 Jun 27;27(5):114. doi: 10.1208/s12248-025-01098-7. PMID 40579609